CLINICAL TRIAL: NCT02354755
Title: The Effect of Temperature on Anesthesia and Surgical Resident's Ability to Perform Clinical and Cognitive Tasks
Status: Completed | Type: Observational
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00858
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia Providers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cold room: Anesthesia providers intraoperatively placed in ambient room temperature of 65 degreees (cold room), completing a 10-minute psychomotor vigilance test (PVT), followed up by a questionnaire on SurveyMonkey
  Interventions: Device: Psychomotor vigilance test (PVT
- Hot room: Anesthesia providers intraoperatively placed in ambient room temperature of 80 degreees (hot room), completing a 10-minute psychomotor vigilance test (PVT), followed up by a questionnaire on SurveyMonkey
  Interventions: Device: Psychomotor vigilance test (PVT
- Control Room: as a control placed Anesthesia providers in ambient room temperature of 75 degreees (neutral room), completing a 10-minute psychomotor vigilance test (PVT), followed up by a questionnaire on SurveyMonkey
  Interventions: Device: Psychomotor vigilance test (PVT

INTERVENTIONS:
Device: Psychomotor vigilance test (PVT — The Psychomotor Vigilance Task Monitor is a hand-held, self-contained system used for repetitive reaction time measurements. The device measures the speed with which subject responds to visual stimulus (by pressing a response button).

SUMMARY:
The purpose of the current study is to examine whether changes in intraoperative ambient temperature has in impact on the clinical performance of the physicians in training which include Anesthesiology and Surgical residents, fellows and certified nurse anesthetists (CRNA). Reaction times will be measured via a 10-minute psychomotor vigilance test (PVT, Ambulatory Monitoring Inc., NY) device.

ELIGIBILITY:
Inclusion Criteria:

* CRNA or surgery or anesthesiology resident fellow in ongoing surgery case

Exclusion Criteria:

* unwilling to participate
* any clinical circumstance that precludes participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians in training (Anesthesiology/surgery residents, fellows and certified registered nurse anesthetists.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Psychomotor vigilance test | 10 minutes
  The Psychomotor Vigilance Task Monitor is a hand-held, self-contained system used for repetitive reaction time measurements. The device measures the speed with which subject responds to visual stimulus (by pressing a response button).

SECONDARY OUTCOMES:
SurveyMonkey Questionairre | 10 minutes